CLINICAL TRIAL: NCT02686788
Title: TMP001 in Relapsing-remitting Multiple Sclerosis: A Multicentre Open, Baseline-controlled Phase IIa Clinical Trial
Brief Title: TMP001 in Relapsing-remitting Multiple Sclerosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dr. Frank Behrens (Other)
Collaborators: SocraMetrics GmbH (Industry)
Responsible Party: Sponsor-Investigator, Dr. Frank Behrens, head of clinical research, Fraunhofer Institute for Translational Medicine and Pharmacology ITMP
Organization: Fraunhofer Institute for Translational Medicine and Pharmacology ITMP (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TMP001_MS
Record Dates: First submitted 2015-10-14; First posted 2016-02-22 (Estimated); Last update posted 2018-11-21 (Actual); Status verified 2018-11

CONDITIONS: Remitting-Relapsing Multiple Sclerosis
Keywords: multiple sclerosis; relapsing remitting; nonsteroidal anti-inflammatory drug; contrast enhancing lesions
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis | interventions — tarenflurbil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- TMP001 (Experimental): 600mg TMP001 as gelatine capsules á 200mg taken orally twice per day for a duration of 24 weeks
  Interventions: Drug: TMP001

INTERVENTIONS:
Drug: TMP001 — 600mg TMP001 as gelatine capsules á 200mg taken orally twice per day for a duration of 24 weeks

SUMMARY:
The purpose of this study is to assess the impact of TMP001 in the treatment of patients with relapsing-remitting multiple sclerosis (RRMS). Therefore the average total number of contrast enhancing lesions (CELs) on brain MRI scans at weeks 12, 16, 20, and 24 during treatment with TMP001 is compared to the average total number of CELs on brain MRI scans at week -4 and baseline in these patients .

Based on promising preclinical results, the investigators assume a comparable effect of TMP001 on reduction of contrast-enhancing lesions as shown for other immunomodulatory substances in recent clinical studies.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 55 years
* Definite diagnosis of RRMS (according to revised McDonald criteria, Polman et al. 2011, Annals of Neurology 69:292-302)
* At least 1 documented relapse during the previous year OR at least 2 documented relapses during the previous 2 years
* At least one contrast-enhancing lesion (CEL) on the screening MRI scan at week (-4)
* EDSS of 0 - 5 (inclusive) at screening (week -4)
* Women of childbearing potential (WOCBP) must use 2 adequate forms of contraception to avoid pregnancy throughout the trial (such as a double barrier method) and for up to 8 weeks after the last dose of TMP001 in such a manner that the risk of pregnancy is minimized
* Written informed consent obtained prior to the initiation of any protocol-required procedures
* Compliance to study procedure and study protocol

Exclusion Criteria:

* History of chronic disease of the immune system other than MS or a known immunodeficiency syndrome
* Clinically severe active infection (e.g., pneumonia, septicaemia) within the 1 month prior to Screening.
* Diagnosis of neuromyelitis optica, clinically isolated syndrome, secondary progressive multiple sclerosis, or primary progressive multiple sclerosis
* History of drug or alcohol abuse within 2 years of inclusion to the study
* Relapse or corticosteroid treatment within 30 days before screening (week -4)
* Interferon-beta, glatiramer acetate, teriflunomide, dimethyl fumarate or fingolimod therapy had to have been stopped 3 or more months before enrolment
* Immunosuppressive medication such as azathioprine or methotrexate, Ciclosporin, cyclophosphamide, mycophenolate mofetil, mitoxantrone or cladribine at any time
* Any previous therapy with alemtuzumab, ocrelizumab, ofatumumab, rituximab, belimumab, natalizumab, total body irradiation, or bone marrow transplantation
* Any investigational drug or placebo within 12 weeks prior to enrolment OR > 5 half-lives prior to screening (week -4), whichever is longer
* Women that are pregnant or currently breast feeding
* Concurrent participation in other clinical trials
* History of, or current diagnosis of, malignancy (including previously treated skin cancer other than successfully treated basal and squamous skin cancer with no evidence of recurrence within 5 years)
* Inability to complete an MRI or contraindications for MRI, including but not limited to claustrophobia, presence of a pacemaker, cochlear implants, ferromagnetic devices or clips, intracranial vascular clips, insulin pumps, or nerve stimulators
* Hypersensitivity to contrast agent (Gadolinium, resp. gadopentetate-dimeglumine)
* Any reason in the discretion of the investigator regarding the safe participation of the patient in the study or for any other reason, the investigator considers the patient inappropriate for participation in the study.
* White blood count (WBC) <3000 mm3 at screening (week -4)Lymphocytes < 800 mm3 at screening (week -4)

Exclusion criteria regarding the study medication:

* Patients with known hypersensitivity to study medication
* Patients who have experienced asthma, urticaria, or allergic-type reactions after taking aspirin or other non-steroidal anti-inflammatory drugs (NSAIDs)
* Patients with a history of peptic ulcer disease and/or gastrointestinal bleeding
* Chronic or acute renal, hepatic or metabolic disorder
* Patients with a history of myocardial infarction, ischemic stroke or known heart failure
* Patients with known thrombophilia or abnormal clinically significant coagulation parameter at screening (week -4)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2015-08; Primary Completion 2018-04 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
Comparison of average total number of contrast enhancing lesions | at week -4, week 0 (baseline), week 4, 8, 12, 16, 20 and 24
  Comparison of average total number of contrast enhancing lesions (CELs) on Brain MRI scans at weeks 4, 8, 12, 16, 20 and 24 as compared to the average total number of CELs on brain MRI scans at week -4 and baseline (BL)

SECONDARY OUTCOMES:
Comparison of average total volume of contrast enhancing lesions | at week -4, week 0 (baseline), week 4, 8, 12, 16, 20 and 24
  Average total volume of CELs (in mm3) on brain MRI scans at week 4,8, 12, 16, 20 and 24 as compared to the average total CEL volume on brain MRI scans at week -4 and BL
Comparison of T2- hyperintense lesions as assessed in MRI | at week 0 (baseline) and week 24
  New or enlarged T2- hyperintense lesions at week 24 as compared to baseline - Number and Characteristics of T2-hyperintense leasion as to be found in MRI Assessment in Comparison between baseline and week 24
Comparison of T1-hypointense lesions as assessed in MRI | at week 0 (baseline) and week 24
  New T1-hypointense lesions at week 24 as compared to baseline as to be found in MRI Assessment in Comparison between baseline and week 24
relapse rate | week -4 until week 24
  Documentation of any replapse during study period to determine the annualised relapse rate
Expanded disability status scale (EDSS) | at week 0 (baseline), week 12 and 24
  EDSS at weeks 12 and 24 as compared to baseline
Assessment of Lipid profile at different time points | at week 0 (baseline), week 12 and 24
  Concentration of a variety of lipids will be determined at weeks 12 and 24 and described in comparison to the lipid profile at baseline
TMP001-concentrations | week 4, 8, 12, 16, 20 and 24
  Assessment of TMP001-concentrations
Pain questionnaire | at week 0 (baseline), week 12 and week 24
  Pain questionnaire at BL, week 12 and week 24

CONTACTS AND LOCATIONS:
Overall Officials: Ulf Ziemann, MD, Principal Investigator — University Department of Neurology Tübingen
Locations (5):
- Germany (5):
  - UKT, Universitätsklinikum Tübingen, Tübingen, Baden-Würtemberg
  - Goethe-Universität Frankfurt am Main, Frankfurt am Main, Hesse
  - Universitätsklinikum Münster, Klinik für Allgemeine Neurologie, Münster, North Rhine-Westphalia
  - Charite- Universitätsmedizin Berlin (Campus Mitte) NeuroCure Clinical Research Center NCRC AG Klinische Neuroimmunologie, Berlin
  - Universitätsklinikum Heidelberg Neurologische Klinik, Heidelberg